CLINICAL TRIAL: NCT01877525
Title: "Resect and Discard" Approach to Diminutive Colonic Polyps: Real World Applicability Amongst Both Academic and Community Gastroenterologists
Brief Title: Resect and Discard Approach to Diminutive Colonic Polyps
Acronym: RD
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201105473
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Benign Polyps of Large Intestine
Keywords: colorectal polyps; resect and discard; endoscopic prediction; histological diagnosis; narrow band imaging
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients in one cohort: Consecutive adult patients undergoing colonoscopy for colorectal cancer screening or routine surveillance indications were prospectively enrolled between October 2011 and October 2012.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — The location, size, and morphology of all lesions detected during colonoscopy were recorded. The size of each identified polyp was visually estimated . All diminutive polyps (defined as ≤5 mm) were endoscopically imaged and histology predictions (adenoma vs. non-adenomatous polyp) were made using HDWL with/without NBI at the discretion of the endoscopist.

SUMMARY:
Resect and discard (RD) is a new paradigm for management of diminutive colorectal polyps wherein histology is determined by real-time endoscopic imaging; polyps are then resected and discarded rather than sent for histopathological review. The aims of this study were to compare the surveillance recommendations between RD and the standard of care where polyps are sent for histopathological review in a mixed setting of academic and community gastroenterologists and to evaluate the diagnostic performance of an RD program for management of diminutive polyps.

DETAILED DESCRIPTION:
Introduction: Diminutive (≤5 mm) colorectal polyps are prevalent in the screening population but have low risk for harboring advanced villous or dysplastic components and for developing into colorectal cancer. "Resect and discard" (RD) is a new paradigm for management of these diminutive polyps wherein histology is determined by real-time endoscopic imaging; polyps are then resected and discarded rather than sent for histopathological review.

Aim: The aim of this study were to compare the surveillance recommendations between RD and the standard of care where polyps are sent for histopathological review in a mixed setting of academic and community gastroenterologists and to evaluate the diagnostic performance of an RD program for management of diminutive polyps.

Methods: This is a prospective, observational study conducted in a single outpatient endoscopy center over 12 months. Screening and surveillance colonoscopies were performed by four academic and two community gastroenterologists. All diminutive polyps (defined as ≤5 mm) were endoscopically imaged and histology predictions (adenoma vs. non-adenomatous polyp) were made using high-definition white light (HDWL) with/without narrow band imaging (NBI) at the discretion of the endoscopist. Diagnostic performance and accordance of recommended surveillance intervals from endoscopic imaging were compared to histopathological review of the polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if diminutive polyps (defined as ≤5 mm) were identified at colonoscopy.

Exclusion Criteria:

* indication other than screening or surveillance
* no diminutive polyps were found
* an optical or histopathological diagnosis of the diminutive polyp could not be made
* the polyp was resected but not retrieved for histopathology
* a synchronous colorectal cancer was identified at the time of the colonoscopy
* polyposis syndrome
* inflammatory bowel disease
* colonoscopies not complete to cecum
* fair or poor bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing colonoscopy for colorectal cancer screening or routine surveillance indications were prospectively enrolled between October 2011 and October 2012. Written informed consent was obtained from all patients.
Sampling Method: Non-Probability Sample
Enrollment: 618 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
concordance of recommended surveillance intervals | 30 days
  concordance of recommended surveillance intervals based on endoscopic optical diagnosis compared to histopathological diagnosis

SECONDARY OUTCOMES:
diagnostic performance | 30 days
  Diagnostic performance [accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)] of adenomatous and non-adenomatous polyps by optical diagnosis using HDWL with/without NBI
  Subgroup analyses were also planned to evaluate diagnostic performance by level of confidence in prediction, type of endoscopist (academic vs. community), and use of NBI.

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Early, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Center for Advanced Medicine, St Louis, Missouri, United States